CLINICAL TRIAL: NCT04726813
Title: An Internet-delivered Intervention for Coping With ADHD in Adulthood - a Randomized Controlled Trial
Brief Title: An Internet-delivered Intervention for Coping With ADHD in Adulthood
Acronym: MyADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Robin Maria Francisca Kenter, Principal investigator, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 203804
Record Dates: First submitted 2021-01-08; First posted 2021-01-27 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: ADHD
Keywords: ADHD; RCT; Internet-delivered intervention; Self-help; Coping
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a self-guided Internet delivered intervention (Experimental): MinADHD: 7 self-help modules.
  Interventions: Behavioral: MyADHD
- Psycho-education (Placebo Comparator): One self-guided psychoeducation module
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: MyADHD — The main goals of the intervention are to help participants with better functioning in daily life; offer strategies that will lead to stress reduction and reduce inattention and improve quality of life.The intervention includes: a short introductory chapter (open to everyone), followed by a start module (goal setting), followed by 6 different themed optional modules. Module content is based on GMT, DBT and CBT techniques and is tailored towards key concerns and difficulties experienced adults with ADHD as informed by previous research (focus-groups, lived experience groups) and experiences from group GMT and DBT.
  Arms: a self-guided Internet delivered intervention
Behavioral: Psychoeducation — Participants in the control condition will be assigned to psychoeducation modules (see Table 2) and will receive restricted access to the platform. They can contact or be contacted if their symptoms levels increases.
  Arms: Psycho-education

SUMMARY:
The primary aim of this study is to examine the efficacy of a self-guided Internet-delivered intervention for coping with ADHD. The secondary aim is to investigate the effects of individual adaptation of the intervention on adherence, satisfaction and clinical outcomes.

DETAILED DESCRIPTION:
ADHD in adulthood, with an estimated prevalence of 2 - 3 %, is associated with challenges in daily life functioning. The availability of evidence-based psychological interventions for adults with ADHD is poor. Interventions delivered over the Internet might help to increase the availability of effective psychological interventions for this group. The primary aim of this study is to examine the efficacy of a self-guided Internet-delivered intervention for coping with ADHD. The secondary aim is to investigate the effects of individual adaptation of the intervention on adherence, satisfaction and clinical outcomes. A minimum of 118 participants with a self-reported ADHD diagnosis will be included in the study. In phase 1 we will conduct a randomized controlled trial with two arms, 1) self-guided Internet-delivered intervention for coping with ADHD (N=59), 2) self-guided online psychoeducation (control group, N= 59), with a 3 month follow-up. After 3 months the second phase of the study starts. In this phase (II) the control group participants will receive an adaptive version of the Internet-delivered intervention. This includes adaptation of the order of the modules to the individual participant needs, with the use of rule-based and machine-learning based adaptation. Clinical outcomes in both phases are inattention, hyperactivity, quality of life and stress. Uptake, usage, adherence and satisfaction will be explored. Repeated measurers are at baseline, weekly during the intervention period, post-intervention and 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with a self-reported diagnosis of ADHD (date, venue and diagnosing physician)
2. Access to and ability to use a computer, smartphone and the Internet.
3. Current problems with organizing daily activity and 17 points of more on at least one of the ASRS subscales
4. Participant are by investigators considered able to follow through the training protocol and take part in measures taken during the study time frame
5. Speaks, writes and reads Norwegian

   Exclusion Criteria:
6. Current self-reported diagnosis of severe psychiatric illness such as borderline or antisocial personality disorder, bipolar disorder, ongoing substance abuse, and/or suicidal ideation assessed with item 9 on the MADRS
7. Participants who are taking prescribed ADHD medication have to be stable on the medication at least four weeks before the study and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
The Adult ADHD Self-Rating Scale (ASRS) | Change in ADHD symptoms at 8 weeks
  The Adult ADHD Self-Rating Scale (ASRS) includes all the 18 symptoms of ADHD included in the diagnostic manual (DSM-5).
Adult ADHD Quality of Life Measure (AAQol) | Change in quality of life at 8 weeks
  The AAQoL has 29 items designed to assess HRQL during the past two weeks among adults with ADHD.

SECONDARY OUTCOMES:
The perceived stress scale (PSS) | Change in stress symptoms at 8 weeks
  The Perceived Stress Scale (PSS) is a widely used psychological instrument for measuring stress.
The Patient Health Questionnaire-9 (PHQ-9) | Change in depression symptoms at 8 weeks
  The Patient Health Questionnaire-9 (PHQ-9: Kroenke et al., 2001) is a self-report tool used to assess the presence and severity of depressive symptoms

OTHER OUTCOMES:
Adherence | immediately after the intervention
  Usage outcomes of interest are attrition and adherence to the intervention.
User satisfaction | immediately after the intervention
  Four open end questions at the end of the modules:
  1. Were there parts of the module that you experienced as helpful and/or supportive?
  2. Were there parts of the module that you experienced as complicated and/or unhelpful?
  3. Would you recommend this module to a friend or a family member with similar difficulties as yourself?
  4. How useful did you find this module? 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Psychology, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kenter RMF, Gjestad R, Lundervold AJ, Nordgreen T. A self-guided internet-delivered intervention for adults with ADHD: Results from a randomized controlled trial. Internet Interv. 2023 Mar 20;32:100614. doi: 10.1016/j.invent.2023.100614. eCollection 2023 Apr. PMID 36969389
- [Derived] Kenter RMF, Lundervold AJ, Nordgreen T. A self-guided Internet-delivered intervention for adults with ADHD: a protocol for a randomized controlled trial. Internet Interv. 2021 Nov 20;26:100485. doi: 10.1016/j.invent.2021.100485. eCollection 2021 Dec. PMID 34877262